CLINICAL TRIAL: NCT03011164
Title: The Influence of Running and Velocity to Kinematic Parameters
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: GuangzhouGH005
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Running; Gait Velocity
Keywords: Running; Gait velocity; Kinematics
MeSH Terms: interventions — Walking; Jogging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- WV 1: The condition of this group will be set as participants walking at 3.5km/h
  Interventions: Procedure: Walk and Run
- WV 2: The condition of this group will be set as participants walking at 4.0km/h
  Interventions: Procedure: Walk and Run
- RV 1: The condition of this group will be set as participants running at 3.5km/h
  Interventions: Procedure: Walk and Run
- RV 2: The condition of this group will be set as participants running at 4.0km/h
  Interventions: Procedure: Walk and Run

INTERVENTIONS:
Procedure: Walk and Run — Once participants are eligible, they will undergo the experimental procedure. Before data collection, they will walk or run on a treadmill in barefoot for ten minutes to adapt the condition. The a gait analysis system will collect the data while they walk or run on the treadmill in barefoot at selected gait speed.

SUMMARY:
Some researches have found that gait posture velocity have influence on kinematic parameters. However, how the gait velocity and posture will influence kinematic parameters remain unclear. In addition to walking, running is one of the most daily activities of people. The purpose of this research is to find out the influence of gait velocity and running to kinematic parameters . To do this, it will provide a reference for future prospective studies or investigations and make us fully understand the impact of gait velocity and running to kinematic parameters of gait.

ELIGIBILITY:
Inclusion Criteria:

i) 20< age < 30. ii) Body mass index < 30. iii) No history of major injury or surgery in lower limbs. iv) No symptoms of lower limbs. v) Physical examination to test the lower limbs to be normal. vi) The habit of moderate exercise (e.g. Jogging )at least once a week for at least 30 minutes

Exclusion Criteria:

i)Body mass index >30. ii) Injury or surgery in hip/knee/ankle. iii) History trauma in the lower limbs (e.g. fracture). iv) Neuropathic disease . v) Muscular disease. vi) Lack ability to finish the procedure physically or mentally. vii) Easy to fall. viii) Any other conditions that can influence gait parameters of the lower limbs.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants will be recruited via university advertisement.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at initial contact. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at loading response. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at mid-stance. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at terminal stance. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at initial swing. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at mid-swing. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at terminal swing. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.
The ranges of motion in the the six-degree-of-motion (6DOF) of the gait. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/ lateral translation, proximal/distal translation.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China

IPD SHARING:
Plan to Share IPD: No